CLINICAL TRIAL: NCT03152539
Title: Development of MRI Protocols and Associated Explorations (EEG, NIRS) in Healthy Volunteers
Acronym: MAP-VS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC12.238
Record Dates: First submitted 2017-04-24; First posted 2017-05-15 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Magnetic Resonance Imaging
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: Methodological development of new MRI approaches
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Development of MRI protocols (Experimental): MRI exam to grade differents interventions for future research
  Interventions: Radiation: MRI
- Development of EEG protocols (Experimental): EEF exam to grade differents interventions for future research
  Interventions: Device: EEG
- Development of NIRS protocols (Experimental): NIRS exam to grade differents interventions for future research
  Interventions: Device: NIRS

INTERVENTIONS:
Radiation: MRI
  Arms: Development of MRI protocols
Device: EEG
  Arms: Development of EEG protocols
Device: NIRS
  Arms: Development of NIRS protocols

SUMMARY:
The main objective of the studies that will be carried out on volunteer patients who have given their consent will be the development and optimization of the sequence parameters or the design of the stimulation paradigms in order to optimize the quality and Relevance of the images realized taking into account anatomical, functional or metabolic parameters. These adjustments will be carried out without interfering with the management of voluntary patients

DETAILED DESCRIPTION:
The pathologies that interest us in these refinements concern mainly the chronic (or sequellar) brain disorders which can be degenerative, developmental or vascular. The patients who will be recruited will be known patients of our Service (University Clinic of Neuroradiology and MRI) that we follow during checks. The type of examination that will be applied to them, between MRI, EEG and NIRS, will be specified in the consent form. These examinations will not be invoiced either to the patient or to the social security, and the related costs will be borne by our Federative Research Structure or sometimes, when these explorations are upstream of a defined research protocol and funded, They will be financed under this protocol.

ELIGIBILITY:
Inclusion Criteria:

* major
* socially insured persons
* given their consent.
* absence of contraindication to the MRI examination

Exclusion Criteria:

* Subjects under the age of 18
* pregnant women
* all other persons referred to in articles L1121-5 to L1121-8 of the CSP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 733 (Actual)
Dates: Start 2012-06-07 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Spatial resolution of new MRI imaging sequences MRI scanning. | Two hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No